CLINICAL TRIAL: NCT02224677
Title: Craniofacial Microsomia: Longitudinal Outcomes in Children Pre-Kindergarten (CLOCK)
Acronym: CLOCK
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Children's Hospital Los Angeles (Other); Children's Hospital of Philadelphia (Other); University of North Carolina (Other); Northwestern University (Other); University of Illinois at Chicago (Other); University of Washington (Other); University of Pittsburgh (Other); New York University (Other)
Responsible Party: Principal Investigator, Carrie Heike, Principal Investigator, Seattle Children's Hospital
Other Study IDs: NIDCR: 13-002-E; R01DE022438-01 (NIH)
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Craniofacial Microsomia; Hemifacial Microsomia; Oculo-Auriculo-Vertebral-Syndrome; Goldenhar Syndrome; Microtia
Keywords: CFM; facial asymmetry; skin tag; facial tag; missing ear; small ear; anotia; microtia; epibulbar dermoid; coloboma; macrostomia; lateral cleft; infant; toddler; baby; neurodevelopment; cognition; socialization
MeSH Terms: conditions — Goldenhar Syndrome; Congenital Microtia; Facial Asymmetry; Coloboma; Macrostomia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Children with Craniofacial Microsomia: 125 children with craniofacial microsomia will be asked to come in for two study visits - when they are about 12 months old and again when they are about 36 months old. Procedures for children at the first visit include: assessment of development, video, photographs, and a hearing evaluation. Procedures for the final study visit include: assessment of development, photographs (2D & 3D), video, saliva sample, hearing evaluation, speech assessment.
- Children without Craniofacial Microsomia: Please note: we are not recruiting this group through ClinicalTrials.gov 100 children without craniofacial microsomia will be asked to come in for two study visits - when they are about 12 months old and again when they are about 36 months old. Procedures for the first visit include: assessment of development, video, and photographs. Procedures for the final study visit include: assessment of development, photographs (2D & 3D), video, and speech assessment.
- Parents of Children with Craniofacial Microsomia: 125-250 parents of children with craniofacial microsomia will be asked to complete three visits - when their child is about 12 months old, 24 months old, and 36 months old. Parents will be asked to complete an interview at the first visit. The second visit consists of a telephone interview where parents will be asked about their child's hearing and health history. At the final study visit, parents will be asked to complete more questionnaires, have their picture taken, and donate saliva.
- Parents of Children without Craniofacial Microsomia: Please note: we are not recruiting this group through ClinicalTrials.gov 100 parents of children without craniofacial microsomia will be asked to complete three visits - when their child is about 12 months old, 24 months old, and 36 months old. Parents will be asked to complete an interview at the first visit. The second visit consists of a telephone interview where parents will be asked about their child's hearing and health history. At the final study visit, parents will be asked to complete questionnaires and an interview.
- Teacher/Day Care Provider: When the children participants are around 36 months old, we will ask parents for permission to contact their child's teacher/day care provider. We would like the teacher/day care provider to fill out a questionnaire.

SUMMARY:
This study is a multi-center, longitudinal cohort study of 125 infants with craniofacial microsomia (CFM) and 100 infants without craniofacial anomalies. Participants will undergo a series of evaluations between 0-3 years of age to comprehensively evaluate the developmental status of infants and toddlers with CFM. This research design will also explore specific pathways by which CFM may lead to certain outcomes. Specifically, the study explores (1) the longitudinal relations between facial asymmetry and emotion-related facial movements and socialization; and (2) associations among ear malformations, hearing and speech deficits and cognitive outcomes. Results of this research will ultimately lead to future investigations that assess new interventions and corresponding changes in current standards of care for children with CFM.

ELIGIBILITY:
We are currently looking to enroll children with craniofacial microsomia through ClinicalTrials.gov

Inclusion Criteria:

Children with Craniofacial Microsomia:

1. Male or female infant participant is between 12 months and 24 months of age, or corrected age (for some infants born prior to their due date).
2. Infant participant has diagnosis of at least one of the following conditions:

   * Microtia
   * Anotia
   * Facial asymmetry AND Preauricular tag(s)
   * Facial asymmetry AND Facial tag(s)
   * Facial asymmetry AND Epibulbar dermoid
   * Facial asymmetry AND Macrostomia (i.e., lateral cleft)
   * Preauricular tag AND Epibulbar dermoid
   * Preauricular tag AND Macrostomia
   * Facial tag AND Epibulbar dermoid
   * Macrostomia AND Epibulbar dermoid
3. Infant participant has been diagnosed by a regional craniofacial team.
4. Legal guardian will provide written parental permission and informed consent prior to participation in study.
5. Legal guardian is willing to comply with all study procedures and be available for the duration of the study through Time 3.

Parents of Children with Craniofacial Microsomia:

* able to provide written consent for study participation,
* willing to comply with all study procedures and
* interested in participating in the entire study through Time 3.

Exclusion Criteria:

Children with Craniofacial Microsomia:

1. Subject is diagnosed with a known syndrome that involves microtia and/or underdevelopment of the jaw (Townes-Brocks, Treacher Collins, branchiootorenal, Nager, or Miller syndromes).
2. Subject has abnormal chromosome studies (karyotype)
3. Subject has a major medical or neurological condition that prevents participation in the study (e.g., cancer, cerebral palsy) at time of recruitment
4. Subject was born before 34 weeks estimated gestational age
5. Anything that would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
6. Sibling already participating in the CLOCK study
7. Subject's consenting parent does not speak English or Spanish

Parents of Children with Craniofacial Microsomia

1. Anything that would preclude the subject's full compliance with or completion of the study.
2. Subject does not speak English or Spanish

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with and without craniofacial microsomia will be drawn from outpatient clinics, medical centers, and local pediatric practices near performance sites and local pediatric practices. Cases will be approached in their first 24 months by either a member of their craniofacial team, a member of the CLOCK study team, or one of their treating providers. Cases may find out about the study through ClinicalTrials.gov. Controls will initially be approached through a treating provider, a member of the CLOCK team, or through an announcement about the study.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental Outcome Measures | T1 study visit (12-14 months of age)
  BSID-III Cognitive Index
Phenotypic Assessments | T1 study visit (12-14 months of age)
  2D photographs and video
Phenotypic Assessments | T2 study visit (~24 months)
  Medical and Surgical History
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  BSID-III Cognitive Index
Neurodevelopmental Outcome Measures | T1 study visit (12-14 months of age)
  BSID-III Fine & Gross Motor
Neurodevelopmental Outcome Measures | T1 study visit (12-14 months of age)
  PLS-V Auditory Comprehension
Neurodevelopmental Outcome Measures | T1 study visit (12-14 months of age)
  PLS-V Expressive Language
Phenotypic Assessments Phenotypic Assessments Phenotypic Assessments | T1 study visit (12-14 months of age)
  3D photographs,
Phenotypic Assessments | T1 study visit (12-14 months of age)
  Medical and Surgical History
Phenotypic Assessments | T1 study visit (12-14 months of age)
  Medical/dental chart abstraction
Phenotypic Assessments | T1 study visit (12-14 months of age)
  IT-MAIS: Auditory Assessment
Phenotypic Assessments | T1 study visit (12-14 months of age)
  OMENS rating from 2D images
Phenotypic Assessments | T1 study visit (12-14 months of age)
  Baby FACS observational protocol
Phenotypic Assessments | T1 study visit (12-14 months of age)
  Clinical Hearing Test
Phenotypic Assessments | T2 study visit (~24 months)
  IT-MAIS: Auditory Assessment
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  BSID-III Fine & Gross Motor
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Brief IQ
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Forward Memory
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Sustained Attention
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Associated Pairs
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Matching
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Leiter-R Picture Context
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  PLS-V Auditory Comprehension
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  PLS-V Expressive Language
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  NEPSY-II Phonological Processing
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  ITSEA Parent
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  ITSEA Teacher
Neurodevelopmental Outcome Measures | T3 study visit (~36 months)
  Goldman-Fristoe Test of Articulation (GFTA-2)
Phenotypic Assessments | T3 study visit (~36 months)
  2D photographs and video
Phenotypic Assessments | T3 study visit (~36 months)
  3D photographs
Phenotypic Assessments | T3 study visit (~36 months)
  Medical and Surgical History
Phenotypic Assessments | T3 study visit (~36 months)
  Medical/dental chart abstraction
Phenotypic Assessments | T3 study visit (~36 months)
  IT-MAIS: Auditory Assessment
Phenotypic Assessments | T3 study visit (~36 months)
  OMENS rating from 2D images
Phenotypic Assessments | T3 study visit (~36 months)
  Hearing Evaluation
Phenotypic Assessments | T3 study visit (~36 months)
  Interview on willingness for future study
Phenotypic Assessments | T3 study visit (~36 months)
  DNA collection (DNA)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Heike, MD, MS, Principal Investigator — Seattle Children's Hospital; Matthew L Speltz, PhD, Principal Investigator — Seattle Children's Hospital
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington